CLINICAL TRIAL: NCT05542485
Title: PLAsma Genomic Testing in Patients With Advanced Non-Small Cell Lung Cancer: The PLAN Study
Acronym: PLAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 22193A01
Record Dates: First submitted 2022-08-22; First posted 2022-09-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be collecting cell free DNA from patients an one time point. These samples will be collected in EDTA tubes and stores for a maximum of 10 years from collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ctDNA liquid biopsy - Roche Avenio Assay — The intervention will involve plasma ctDNA testing for patients with a radiological suspicion for newly diagnosed advanced NSCLC

SUMMARY:
This is a multi-centre, prospective, translational study investigating the use of plasma genotyping for initial genomic testing in newly diagnosed advanced/locally advanced non-squamous NSCLC.

In this study, patients will have a plasma genotyping assay completed following confirmation of suspected diagnosis of non-squamous NSCLC at institutional Rapid Access Lung Cancer Clinics (RALCC), alongside standard tissue-based biopsy and genotyping.

DETAILED DESCRIPTION:
Background Genomic Testing in Non-Small Cell Lung Cancer Tissue genotyping of therapeutically actionable alterations is a standard diagnostic requirement for patients with advanced non-squamous NSCLC. Tissue genotyping represents a gold standard, with both a sensitivity and specificity for identifying common genomic alterations of >90%. NSCLC represents a genomically diverse cancer. Detection of genomic alterations has progressed over the past decade, now including detection of mutations such as KRAS, EGFR, ERBB2, BRAF, MET and fusions including ALK, ROS1, NTRK and RET genes, as well as co-occurring mutations on tissue samples. The ability to detect these mutations has led to discovery of molecularly defined subsets of NSCLC, and a rapid growth in the development of targeted therapies. Actionable oncogenic driver mutations, which lead to uncontrolled cell growth, are detected in up to 64% of lung adenocarcinomas. The most commonly observed oncogenic driver mutation in NSCLC is KRAS, observed in up to 30% of cases, which has led to the development of agents such as sotorasib and adagrasib to target KRAS G12C mutations after failed first line systemic therapies. The development of EGFR tyrosine kinase inhibitors (TKIs) such as osimertinib, gefitinib or erlotinib, and ALK directed therapy with crizotinib, alectinib and ceritinib has led to significant improvement in survival in patients with NSCLC over the past decade, and shifted the focus to developing improved detection methods of these mutations for first-line targeted therapy. Each actionable mutation detected has led to the rapid expansion of available therapeutic options beyond those mentioned above and changed the landscape of lung cancer treatment.

The majority of NSCLC is diagnosed at an advanced stage (stage III or IV), and it is often diagnosed with a core biopsy or cytology specimens. Oncology and pathology societies recommend that molecular testing turnaround times not exceed 10 working days yet up to 30% of these specimens are insufficient to allow for tissue genotyping necessitating repeat biopsy. Patients may thus clinically deteriorate while waiting for genomic test results. In those patients who have insufficient samples on initial biopsy and require repeat intervention, this can prolong the time from diagnosis to treatment by more than 28 days. The methods by which these mutations are detected are continually evolving, including DNA sequencing, DNA allele-specific testing, RNA sequencing, fluorescent in situ hybridization (FISH) to detect fusion genes, and next generation sequencing (NGS). Both DNA and RNA sequencing have been shown to detect actionable mutations, but certain large panels can miss small exon skipping or fusion alterations, and thus a sequential approach may be warranted. In certain mutations, RNA sequencing can detect a higher proportion of MET exon 14 skipping. Frequently a hotspot panel is used to detect a range of commonly occurring mutations, and if negative for these mutations, single gene sequencing can be done for less common mutations, which is time consuming and can further delay treatment. NGS has become the gold-standard method to detect actionable mutations, and was recommended by the European Society for Medical Oncology (ESMO) in 2020 in advanced non-squamous NSCLC, as well as in other malignancies including cholangiocarcinoma, prostate and ovarian cancers. NGS provides a broader test platform, and can assess many more potential gene alterations. The MOSCATO trial assessed the use of high throughput genomic analyses including NGS and showed improved outcomes in advanced cancer. Specifically in NSCLC, NGS has shown significantly improved outcomes, by identifying patients who will derive the greatest benefit from targeted therapies, therefore reducing toxicity related to ineffective therapies with certain mutations.

Plasma genotyping in non-small cell lung cancer Plasma genotyping, or 'liquid biopsy,' is a relatively new technology in which circulating tumour DNA (ctDNA), shed into the bloodstream by tumours, is detectable by next generation sequencing. This technology, while associated with a slightly lower sensitivity (80%), has >96% concordance for tissue testing of EGFR, ALK, ROS1 and BRAF mutations. In addition, the median turnaround time is just 7-10 days, without the associated risks and costs of invasive biopsy. Recent studies have shown the dynamic nature of tumour cells including the development of resistance mechanisms in EGFR-mutated tumours. As such, many cancer centres, including some based in Ireland, have used liquid biopsy as a means of surveillance for these resistance mechanisms over time rather than submitting a patient to multiple repeat biopsies. More recently many centres in North America and Europe have utilised liquid biopsy for assessing genomic alterations for targeted therapies in lung cancer upfront at the time of tissue sampling, thereby reducing the time to treatment commencement. This approach is supported by several high-level papers, including the NILE study, a prospective study of 282 patients with advanced untreated NSCLC that showed concordance between tissue and plasma genotyping and a significantly faster turnaround time from 15 to 9 days. A single centre study in the USA showed that concurrent plasma and tissue testing in NSCLC increased the detection of actionable mutations by 15%, and hence increased the number of patients receiving targeted therapies.

As well as the oft needed requirement for repeat biopsy due to a lack of tumour tissue for NGS, patients with advanced NSCLC often have a poor ECOG performance status which can limit the possibility of primary invasive procedures or repeat tissue sampling, and in some cases, the location of the tumour site may not be amenable to biopsy. In the event that tissue can be retrieved by invasive procedure, storage of these samples, for example with formalin fixation, can lead to false positive results on next generation sequencing. Invasive sampling is often associated with high cost, due to the number of clinicians, and supportive staff available. Blood sampling is minimally invasive during the initial diagnosis, bypasses the time required to schedule bronchoscopy or radiologically-guided biopsies and allows immediate processing of samples. Although the use of plasma genotyping has expanded in recent years, it is likely that it would remain an additional tool alongside tissue genotyping, as tissue samples can provide morphology and elucidate primary sites of disease.

Rationale We propose this study to evaluate the feasibility of a plasma-based circulating tumour DNA mutation testing pathway using NGS and initiated at the Rapid Access Lung Cancer Clinic (RALCC) for patients with suspected NSCLC in Ireland. This proof of principle initiative aims to establish a robust patient pathway for systematic somatic mutation testing in patients with NSCLC in Ireland using plasma-based testing. Plasma will be tested for circulating tumour DNA mutations using a validated NGS-based assay, at one of two testing laboratories in Ireland. Proving feasibility through a clinical trial in Ireland is crucial to inform successful applications for authorisation of liquid biopsy to the National Clinical Cancer Programme and to inform clinical trials that aim to identify novel therapies for Irish patients. We believe an upfront plasma-based pathway would lower median turnaround time in the Irish context. Liquid biopsy testing of patients in the RALCC for tumour mutations should ensure that more patients have access to precision medical therapies. Moreover, this approach is likely to significantly improve the identification rate of patients with NSCLC actionable genomic alterations, with resultant benefits for these patients in terms of cancer treatment. This study will also report on the currently unknown frequency, characteristics, disease course, and treatment patterns of somatic mutations in an Irish population with NSCLC.

Hypothesis Upfront plasma-based tumour genotyping of patients with advanced NSCLC with the goal of guiding treatment selection is feasible to implement and will reduce the time to treatment compared with tissue genotyping.

Planned Analysis This proof of principle initiative aims to establish a robust patient pathway for systematic somatic mutation testing in patients with NSCLC in Ireland using plasma-based testing. Plasma will be tested for circulating tumour DNA mutations using a validated NGS-based assay, at one of two testing laboratories in Ireland. The Cancer Molecular Diagnostics (CMD) laboratory at St James's Hospital will perform the tumour test on using an in- house Roche AVENIO ctDNA Expanded panel (Basel, Switzerland). The Histopathology Department at Beaumont Hospital will use an in-house Roche AVENIO ctDNA Expanded panel on the Illumina MiSeq NGS platform (California, USA). Both assays will be validated on a training tumour set. In parallel to ctDNA testing, tumour biopsy tissue testing will be carried out as per standard of care. Liquid biopsy results will be reviewed by the treating clinician for treatment decision purposes however the treatment decision will remain at the discretion of the treating medical oncologist.

It is recognised that liquid and tissue biopsy both have an excellent specificity (>95%). However, liquid biopsy may have a lower sensitivity in the region of 80%. As such, there may be genomic alterations identified on tissue biopsy not identified on liquid biopsy and less likely - vice-versa. In that event, the genotyping which has reported a genomic alteration will be considered the most clinically relevant results as the likelihood of a false positive result is very low (< 5%). However, final treatment decision will remain at the discretion at the treating medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

1. Radiological suspicion of advanced or locally advanced non-small cell lung cancer
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Ability of subject to understand and the willingness to sign a written informed consent document.

   Second arm additional criteria
5. Planned for systemic treatment with either single agent immunotherapy (IT) or combination chemotherapy/IT
6. No prior systemic therapy for advanced NSCLC

Exclusion Criteria:

1. Squamous cell subtype NSCLC histology
2. Small cell carcinoma histology
3. Patients who have received systemic anti-cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with a radiological suspicion of a new diagnosis of stage IV NSCLC will be considered for inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time difference in days between the time of report of plsama genotyping result (next gen sequencing on ctDNA) versus the time to reporting of the tissue genotyping result (from a tissue biopsy sample) | 1 month
  This will be calculated as such ; Time difference = (Number of days from the time of tissue biopsy to reporting of genomic result) - (Number of days from the time of liquid biopsy to result). The liquid biopsy and tissue biopsy will be completed on the same day.

SECONDARY OUTCOMES:
• Time difference between plasma genotyping and tissue genotyping initiation of treatment (time defined by primary endpoint) analysed as pairs with liquid and tissue biopsy | 1 month
• Rate of genomic alterations identified by plasma genotyping assay. | 1 month
• Pattern of actionable genomic mutations alterations on plasma genotyping assay. | 1 month

CONTACTS AND LOCATIONS:
Locations (3):
- Ireland (3):
  - Beaumont Hospital, Dublin
  - St. James' Hospital, Dublin
  - University Hospital Limerick, Limerick

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Reilly D, O'Grady A, Hayes C, Piggott L, Keane R, Fitzpatrick OM, Conroy M, Aretz NK, Synnott D, Dillon R, Dowling GP, Ryan DJ, O'Brien E, Morgan R, Breathnach O, Grogan L, Morris P, Greally M, Teo MY, Murphy A, Ryan G, Counihan I, Ryan C, Barrett H, O'Shea AM, Cuffe S, Korpanty G, Prior L, Barr MP, Finn S, O'Brien C, McCarron S, Cummins R, Toomey S, Dowling CM, Glavey S, Hennessy BT, Sorensen J, Bennett K, Nadarajan P, Doyle B, Naidoo J. Clinical benefit and cost of plasma-first next-generation sequencing in patients with newly diagnosed advanced non-small cell lung cancer in Ireland: The PLAN study. Eur J Cancer. 2025 Jul 25;225:115582. doi: 10.1016/j.ejca.2025.115582. Epub 2025 Jun 17. PMID 40578048